CLINICAL TRIAL: NCT04167813
Title: Trial of Ondansetron as a Parkinson's HAllucinations Treatment
Acronym: TOP HAT
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University College, London (Other)
Collaborators: MODEPHARMA Limited (Unknown); Parkinson's UK (Other); PRIMENT (Unknown); SEALED ENVELOPE (Unknown); Wasdell Packaging Ltd (Unknown); Custom Pharmaceuticals Limited (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 17/0909
Record Dates: First submitted 2019-11-15; First posted 2019-11-19 (Actual); Last update posted 2024-03-27 (Actual); Status verified 2024-03

CONDITIONS: Parkinson's Hallucinations; Dementia With Lewy Bodies
MeSH Terms: conditions — Lewy Body Disease | interventions — Ondansetron; Tablets

STUDY DESIGN:
Intervention Model Description: TOPHAT is a double blind, individually randomized, placebo-controlled, parallel group, flexible dose trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Treatment (Active Comparator): Participants randomised to the active treatment arm will take 8-24mg/day of ondansetron.
  Interventions: Drug: Ondansetron 8mg or matched placebo tablets
- Matched placebo (Placebo Comparator): Participants randomised to the placebo treatment arm will take matched placebo, administered as tablets.
  Interventions: Drug: Ondansetron 8mg or matched placebo tablets

INTERVENTIONS:
Drug: Ondansetron 8mg or matched placebo tablets — Participants will take one tablet daily in weeks 1 and 2, two tablets daily in weeks 3 and 4 and 3 tablets daily in weeks 5 and 6.
  Dose escalation will be guided by tolerability, through telephone safety monitoring prior to each dose increase
  Other Names: Tablet, film coated

SUMMARY:
TOPHAT (Trial of Ondansetron as a Parkinson's HAllucinations Treatment) is a double blind, individually randomized, placebo-controlled, parallel group, flexible dose trial of ondansetron (8-24mg/day) as a treatment for Parkinson's hallucinations, with a 12-week primary outcome and follow-up to 24 weeks.

DETAILED DESCRIPTION:
This study investigates whether ondansetron, a drug used to treat post-operative sickness, has a meaningful treatment effect on Parkinson's hallucinations, and whether the drug is safe and cost effective for use in the NHS. We will compare ondansetron to placebo (a tablet that looks identical but contains no drug) over 12 weeks treatment, with follow up (once treatment ends) for a further 12 weeks. Assessments of symptoms will be carried out during treatment (after 6 and 12 weeks), and once treatment ends (18, 24 weeks), to measure hallucinations, delusions (false beliefs), Parkinson's symptoms (tremor, anxiety, sleep disturbance), memory, quality of life, possible side-effects such as constipation and headache, and the proportion of people who drop out due to side effects, or require additional treatment for their hallucinations. Blood drug concentration (measured after 6 and 12 weeks) will provide information on how quickly the drug is cleared from the body, and how this relates to treatment effects and side-effects, to guide future prescribing in people with Parkinson's. Based on knowledge of the average hallucinations scores in previous Parkinson's treatment studies, 306 people will be needed for the study to detect a meaningful treatment effect. The study will run for 4 years and involves a series of linked stages: (1) Trial set up across 20-30 UK centres; (2) Recruitment over 2 years; (3) Completion of follow up; and analysis, publication and dissemination of results.

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged over 18 years.
2. Meet MDS criteria for Parkinson's disease or revised criteria for DLB.
3. Score of 3 or more on the SAPS-H visual hallucinations item, indicating the presence of visual hallucinations at least weekly in the previous month.
4. Score of 3 or more on SAPS-H global rating, indicating moderate symptom severity.
5. Score of 4 or more on CGI-S, indicating moderate symptom severity.
6. On a stable dose of anti-Parkinson's medication, cholinesterase inhibitor or memantine for at least 28 days.
7. Capacity to give informed consent or, if lacking, legal representative able to give consent.
8. Pre-menopausal women, and men whose partners are of child bearing potential will agree to use effective contraception. 9) If treated with an antipsychotic drug at the time of enrolment, can still participate, provided the drug is stopped the day before trial medication is commenced.

   -

Exclusion Criteria:

1. Bradycardia (<50 bpm) (rescreen if reversible).
2. Congenital long QTc syndrome or presence of clinically significant prolongation of QTc (>460 ms for men or >470 ms for women) on ECG screening.
3. Severe hepatic failure (bilirubin >50 micromole/L)
4. Prescribed apomorphine (if apomorphine is discontinued, rescreen once stable on an alternative anti-Parkinson's treatment).
5. Prescribed tropisetron, granisetron, dolasetron.
6. History of hypersensitivity to ondansetron and its excipients (or those of placebo) or drugs listed in 5).
7. Participation in another Clinical Trial of an Investigational Medicinal Product (IMP) in the previous 28 days.

   -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2024-08-30 (Estimated); Study Completion 2024-08-30 (Estimated)

PRIMARY OUTCOMES:
Hallucinations | 12 weeks
  Scale for Assessment of Positive Symptoms-Hallucinations (0-35 points, higher scores indicate greater severity of hallucinations

SECONDARY OUTCOMES:
Delusions | 2, 4, 6, 12, 18, 24 weeks
  Scale for Assessment of Positive Symptoms-Delusions (0-65 points, higher scores indicate greater symptom severity
Safety and tolerability | 2, 4, 6, 12, 18, 24 weeks
  Number of Participants With Treatment-Related Adverse Events
Health related quality of life | 6, 12, 18, 24 weeks
  EQ-5D-5L
Cost effectiveness | 2, 4, 6, 12, 18, 24 weeks
  Health and social service utilisation
Pharmacokinetics, plasma concentrations of the study drug | 6, 12 weeks
  Measured using a validated HPLC/MS assay
Hallucinations | 2, 4, 6, 18, 24 weeks
  Scale for Assessment of Positive Symptoms-Hallucinations (0-35 points, higher scores indicate greater severity of hallucinations
Global illness severity | 2, 4, 6, 12, 18, 24 weeks
  Clinical Global Impression of Severity Scale (1-7, higher scores indicate greater severity)
Non-motor symptoms | 2,4,6,12,18,24 weeks
  Non-motor symptoms scale (0-120, higher scores indicate greater severity
Cognition | 12 weeks
  Standardised Mini-Mental State Examination (0-30, higher scores indicate better performance)
Hallucinations | 6, 12 weeks
  University of Miami Parkinson's disease Hallucinations Questionnaire (0-15, where higher scores indicate greater symptom severity)
Feasibility and Acceptability of Video Consultation | baseline, 6 and 12 weeks
  The feasibility of video consultation will be measured at baseline, 6 and 12 weeks by the proportion of participants who were able to successfully attend on at least one occasion, the proportion who successfully attended all three assessments, and a Satisfaction questionnaire that allows both quantitative and qualitative information to be collected.

CONTACTS AND LOCATIONS:
Locations (23):
- United Kingdom (23):
  - Grampian, Aberdeen
  - Betsi Cadwaladr, Bangor
  - Pennine, Bury
  - Addenbrookes, Cambridge
  - Dartford, Dartford
  - Tayside, Dundee
  - Glasgow, Glasgow
  - Barking, London
  - Bart's Health, London
  - Imperial College NHS, London
  - Lewisham, London
  - Luton & Dunstable, London
  - UCLH NHS foundation trust, London
  - Newcstle, Newcastle
  - Anuerin Bevan, Newport
  - Northumbria, North Shields
  - Oxford, Oxford
  - North West Anglia, Peterborough
  - Dorset, Poole
  - Cornwall, Redruth
  - Salford, Salford
  - North Midlands, Stoke
  - Sherwood Forest, Sutton in Ashfield

IPD SHARING:
Plan to Share IPD: No